CLINICAL TRIAL: NCT03069352
Title: A Randomized, Double-Blind, Placebo Controlled Phase 3 Study of Venetoclax Co-Administered With Low Dose Cytarabine Versus Low Dose Cytarabine in Treatment Naïve Patients With Acute Myeloid Leukemia Who Are Ineligible for Intensive Chemotherapy
Brief Title: A Study of Venetoclax in Combination With Low Dose Cytarabine Versus Low Dose Cytarabine Alone in Treatment Naive Patients With Acute Myeloid Leukemia Who Are Ineligible for Intensive Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-043; 2016-003900-30 (EudraCT Number); 2024-513630-37-00 (Other: EU CT)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia; Leukemia; Treatment naïve; Venetoclax; Cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — venetoclax; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Venetoclax + Low Dose Cytarabine (LDAC) (Experimental): Venetoclax 600 mg orally every day (QD) plus LDAC 20 mg/m² subcutaneously on Days 1 to 10 of each 28-day cycle.
  Interventions: Drug: Venetoclax; Drug: Cytarabine
- Placebo + LDAC (Placebo Comparator): Matching placebo to venetoclax orally QD plus LDAC 20 mg/m² subcutaneously on Days 1 to 10 of each 28-day cycle.
  Interventions: Drug: Placebo; Drug: Cytarabine

INTERVENTIONS:
Drug: Placebo — tablet
  Arms: Placebo + LDAC
Drug: Venetoclax — tablet
  Other Names: ABT-199; Venclexta
  Arms: Venetoclax + Low Dose Cytarabine (LDAC)
Drug: Cytarabine — Subcutaneous injection
  Other Names: Cytosar-U; Ara-C; Arabinosylcytosine

SUMMARY:
The primary objective of this study is to evaluate if venetoclax when co administered with low-dose cytarabine (LDAC) improves overall survival (OS) versus LDAC and placebo, in treatment-naïve patients with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is an aggressive and rare cancer of myeloid cells (a white blood cell responsible for fighting infections). Successful treatment of AML is dependent on what subtype of AML the patient has, and the age of the patient when diagnosed.

Venetoclax is an experimental drug that kills cancer cells by blocking a protein (part of a cell) that allows cancer cells to stay alive. This study is designed to see if adding venetoclax to cytarabine works better than cytarabine on its own.

This is a Phase 3, randomized, double-blind (treatment unknown to patients and doctors), placebo-controlled, multicenter study in patients with AML who are 18 or more years old and have not been treated before. Patients who take part in this study should not be suitable for intensive induction chemotherapy (usual starting treatment). Abbvie is funding this study which will take place at approximately 125 hospitals globally. In this study, 2/3 of patients will receive venetoclax every day with cytarabine and the remaining 1/3 will receive placebo (dummy) tablets with cytarabine.

Participants will continue to have study visits and receive treatment for as long as they are having a clinical benefit. The effect of the treatment on AML will be checked by taking blood, bone marrow, scans, measuring side effects and by completing health questionnaires. Blood and bone marrow tests will be completed to see why some people respond better than others.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have histological confirmation of acute myeloid leukemia (AML) by World Health Organization criteria, be ineligible for intensive induction chemotherapy and either be:

   * ≥ 75 years of age OR
   * ≥ 18 to 74 years of age and fulfill at least one criteria associated with lack of fitness for intensive induction chemotherapy:

     * Eastern Cooperative Oncology Group (ECOG) performance status of 2 - 3
     * Cardiac history of congestive heart failure (CHF) requiring treatment or ejection fraction ≤ 50% or chronic stable angina
     * Diffusing capacity of the lung for carbon monoxide (DLCO) ≤ 65% or forced expiratory volume in 1 second (FEV1) ≤ 65%
     * Creatinine clearance ≥ 30 mL/min to < 45 ml/min
     * Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 × upper limit of normal (ULN)
     * Other comorbidity that the physician judges to be incompatible with conventional intensive chemotherapy which must be reviewed and approved by the study medical monitor before study enrollment
2. Participant must have an ECOG performance status:

   * of 0 to 2 for subjects ≥ 75 years of age OR
   * of 0 to 3 for subjects between 18 to 74 years of age
3. Participant must have a projected life expectancy of at least 12 weeks.
4. Participant must have adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24-hour urine collection.
5. Participant must have adequate liver function as demonstrated by:

   * aspartate aminotransferase (AST) ≤ 3.0 × ULN*
   * alanine aminotransferase (ALT) ≤ 3.0 × ULN*
   * bilirubin ≤ 1.5 × ULN*

     * Subjects who are < 75 years of age may have bilirubin of ≤ 3.0 × ULN

   (*Unless considered to be due to leukemic organ involvement.)
6. Female participants must be either postmenopausal defined as:

   * Age > 55 years with no menses for 12 or more months without an alternative medical cause.
   * Age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND a follicle-stimulating hormone (FSH) level > 40 IU/L.

   OR
   * Permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

   OR
   * A woman of childbearing potential (WOCBP) practicing at least one protocol specified method of birth control starting at Study Day 1 through at least 180 days after the last dose of study drug.
7. Male participants who are sexually active, must agree, from Study Day 1 through at least 180 days after the last dose of study drug, to practice protocol specified methods of contraception. Male subjects must agree to refrain from sperm donation from initial study drug administration through at least 180 days after the last dose of study drug.
8. Females of childbearing potential must have negative results for pregnancy test performed:

   * At Screening with a serum sample obtained within 14 days prior to the first study drug administration, and
   * Prior to dosing with urine sample obtained on Cycle 1 Day 1, if it has been > 7 days since obtaining the serum pregnancy test results.
   * Subjects with borderline pregnancy tests at Screening must have a serum pregnancy test ≥ 3 days later to document continued lack of a positive result.
9. Participant must voluntarily sign and date an informed consent form, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. Participant has received any prior treatment for AML with the exception of hydroxyurea, allowed through the first cycle of study treatment. Note: Prior treatment for myelodysplastic syndrome is allowed except for use of cytarabine.
2. Participant had an antecedent myeloproliferative neoplasm (MPN) including myelofibrosis, essential thrombocytosis, polycythemia vera, or chronic myelogenous leukemia (CML) with or without BCR-ABL 1 translocation and AML with BCR-ABL 1 translocation.
3. Participants that have acute promyelocytic leukemia (APL).
4. Participant has known central nervous system (CNS) involvement with AML.
5. Participant has known human immunodeficiency virus (HIV) infection (due to potential drug-drug interactions between antiretroviral medications and venetoclax). HIV testing will be performed at Screening, if required per local guidelines or institutional standards.
6. Participant is known to be positive for hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Inactive hepatitis carrier status or low viral hepatitis titer on antivirals (non-exclusionary medications) are not excluded.
7. Participant has received strong or moderate cytochrome P450 3A4 (CYP3A) inducers 7 days prior to the initiation of study treatment.

   * Chinese subjects are excluded from receiving strong and/or moderate CYP3A inhibitors 7 days prior to the initiation of study treatment through the end of intensive pharmacokinetic (PK) collection (24 hours post dose on Cycle 1 Day 10).
8. Participant has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or star fruit within 3 days prior to the initiation of study treatment.
9. Participant has cardiovascular disability status of New York Heart Association Class > 2. Class 2 is defined as cardiac disease which subjects are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or angina pain. Class 3 is defined as cardiac disease which subjects are comfortable at rest but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class 4 is defined as cardiac disease which subjects have an inability to carry on any physical activity without discomfort, symptoms of heart failure at rest, and if any physical activity is undertaken then discomfort increases.
10. Participant has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, any other medical condition or known hypersensitivity to any of the study medications including excipients of LDAC that in the opinion of the investigator would adversely affect his/her participating in this study.
11. Participant has a malabsorption syndrome or other condition that precludes enteral route of administration.
12. Participant exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial or fungal).
13. Participant has a history of other malignancies prior to study entry, with the exception of:

    * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
    * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
    * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
14. Participant has a white blood cell count > 25 × 10^9/L. (Note: hydroxyurea administration or leukapheresis is permitted to meet this criterion).
15. Previous treatment with venetoclax and/or current participation in any other research study with investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2025-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (109):
- United States (6):
  - H. Lee Moffit Cancer Center /ID# 164273, Tampa, Florida
  - Norton Cancer Institute /ID# 158998, Louisville, Kentucky
  - Univ of Pittsburgh Med Ctr /ID# 158997, Pittsburgh, Pennsylvania
  - Univ TX, MD Anderson /ID# 159678, Houston, Texas
  - Swedish Medical Center /ID# 161280, Seattle, Washington
  - Gundersen Health System /ID# 164272, La Crosse, Wisconsin
- Argentina (2):
  - Cemic /Id# 159676, Buenos Aires
  - Sanatorio Allende /ID# 159675, Córdoba
- Australia (4):
  - Calvary Mater Newcastle /ID# 160123, Waratah, New South Wales
  - Westmead Hospital /ID# 160121, Westmead, New South Wales
  - Alfred Hospital /ID# 160125, Melbourne, Victoria
  - Box Hill Hospital /ID# 162920, Melbourne, Victoria
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen /ID# 159566, Edegem, Antwerpen
  - Cliniques Universitaires Saint Luc /ID# 159567, Woluwe-Saint-Lambert, Brussels Capital
- Brazil (4):
  - Centro de Pesquisas Oncologicas /ID# 163567, Florianópolis, Santa Catarina
  - Hospital de Cancer de Barretos /ID# 163568, Barretos, São Paulo
  - Hospital do Cancer Mae de Deus /ID# 163416, Porto Alegre
  - Casa de Saúde Santa Marcelina /ID# 163413, São Paulo
- Canada (4):
  - University of Alberta Hospital /ID# 159646, Edmonton, Alberta
  - CISSS de la Monteregie /ID# 159782, Greenfield Park, Quebec
  - Hospital Maisonneuve-Rosemont /ID# 159780, Montreal, Quebec
  - Hopital Sacre Coeur Montreal /ID# 160982, Montreal, Quebec
- China (11):
  - Fujian Medical Univ Union Hosp /ID# 167321, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University /ID# 170147, Guangzhou, Guangdong
  - Jiangsu Province People's Hospital /ID# 167511, Nanjing, Jiangsu
  - The First Hosp of Jilin Univ /ID# 167512, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong /ID# 167325, Shanghai, Shanghai Municipality
  - West China Hospital /ID# 167514, Chengdu, Sichuan
  - Blood disease hosp of Chinese Academy of Med Sciences(Institute of Hematology) /ID# 167509, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital,College of Medicine, Zhejiang University /ID# 167324, Hangzhou, Zhejiang
  - Qilu Hospital of Shandong Univ /ID# 167507, Jinan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 167515, Wuhan
  - Henan Cancer Hospital /ID# 167327, Zhengzhou, Henan
- Czechia (3):
  - Fakultni Nemocnice Brno /ID# 159247, Brno
  - Univ Hosp Ostrava-Poruba /ID# 159246, Ostrava
  - Fakult Nem Kralovske Vinohrady /ID# 159248, Prague
- France (5):
  - Centre Hospitalier Lyon Sud /ID# 159705, Pierre-Bénite, Rhone
  - Centre Hospitalier Le Mans /ID# 159702, Le Mans, Sarthe
  - Centre Hospitalier de la Cote /ID# 159697, Bayonne
  - CHU Bordeaux /ID# 159704, Pessac
  - CHU De Nancy /ID# 159700, Vandœuvre-lès-Nancy
- Germany (3):
  - Schwarzwald-Baar-Klinikum /ID# 159571, Villingen-Schwenningen, Baden-Wurttemberg
  - Vivantes Klinikum Am Urban /ID# 159569, Berlin
  - Universitaetsklinikum Hamburg /ID# 161760, Hamburg
- Greece (5):
  - General Hospital of Athens Laiko /ID# 157870, Athens, Attica
  - Gen Univ Hosp Alexandroupolis /ID# 157868, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 157869, Athens
  - University Gen Hosp of Patra /ID# 157871, Pátrai
  - General Hospital of Thessaloniki George Papanikolaou /ID# 157867, Thessaloniki
- Hungary (7):
  - Dél-pesti Centrumkórház- Országos Hematológiai és Infektológiai Intézet /ID# 159127, Budapest IX, Budapest
  - Pecsi Tudomanyegyetem /ID# 163161, Pécs, Pecs
  - Semmelweis Egyetem I. Belklini /ID# 158180, Budapest
  - Debreceni Egyetem Klinikai Koz /ID# 158178, Debrecen
  - Petz Aladar Megyei Oktato Korh /ID# 161739, Győr
  - Kaposi Mor Oktato Korhaz /ID# 158175, Kaposvár
  - Bacs-Kiskun Megyei Korhaz /ID# 160973, Kecskemét
- Ireland (4):
  - St. James's Hospital /ID# 162730, Dublin, Dublin
  - Beaumont Hospital /ID# 162733, Dublin
  - University Hospital Galway /ID# 162734, Galway
  - University Hospital Limerick /ID# 162735, Limerick
- Japan (18):
  - University of Fukui Hospital /ID# 159770, Yoshida-gun, Fukui
  - Kyushu University Hospital /ID# 159688, Fukuoka, Fukuoka
  - Gunmaken Saiseikai Maebashi Hospital /ID# 160597, Maebashi, Gunma
  - National Hospital Organization Mito Medical Center /ID# 162988, Higashi Ibaraki-gun, Ibaraki
  - Kyoto Prefect Univ Med /ID# 160101, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 161151, Sendai, Miyagi
  - Nagasaki University Hospital /ID# 160233, Nagasaki, Nagasaki
  - Osaka City University Hospital /ID# 159722, Osaka, Osaka
  - Kinki University -Osakasayama Campus /ID# 160777, Osakasayama-shi, Osaka
  - Tokyo Metropolitan Komagome Hospital /ID# 160759, Bunkyo-ku, Tokyo
  - Tokyo Jikei Daisan Hospital /ID# 159769, Komae-shi, Tokyo
  - NTT Medical Center Tokyo /ID# 160678, Shinagawa-ku, Tokyo
  - Yamagata University Hospital /ID# 161223, Yamagata, Yamagata
  - Akita University Hospital /ID# 160602, Akita
  - Saitama Med Univ Int Med Ctr /ID# 161308, Hidaka
  - NHO Nagoya Medical Center /ID# 159768, Nagoya
  - Dokkyo Medical University Hosp /ID# 159650, Shimotsuga
  - Juntendo University Hospital /ID# 159781, Tokyo
- Mexico (3):
  - Instituto Nacional de Cancerol /ID# 159269, Mexico City, Mexico City
  - Centro de Invest Clin Chapulte /ID# 162625, Morelia, Michoacán
  - Hosp. Univ. Dr. Jose E. Gonz /ID# 159268, Monterrey, Nuevo León
- New Zealand (2):
  - North Shore Hospital /ID# 160132, Auckland
  - Middlemore Clinical Trials /ID# 160131, Auckland
- Norway (2):
  - Haukeland University Hospital /ID# 165630, Bergen, Hordaland
  - Sykehuset Ostfold Kalnes /ID# 165632, Grålum
- VA Caribbean Healthcare System /ID# 158999, San Juan, Puerto Rico
- Russia (9):
  - Kemerovo Regional Clinical Hospital n.a. S.V. Belyaev /ID# 162991, Kemerovo, Kemerovo Oblast
  - Nizhniy Novgorod regional clinical hospital named N. A. Semashko /ID# 163186, Nizhny Novgorod, Nizhny Novgorod Oblast
  - State Institution of Health of the Ryazan Regional Clinical Hospital /ID# 163126, Ryazan, Ryazan Oblast
  - City Clinical Hospital Botkina /ID# 164086, Moscow
  - Almazov North-West Federal Med /ID# 162170, Saint Petersburg
  - Saint Petersburg State Institu /ID# 162171, Saint Petersburg
  - Samara State Medical Universit /ID# 164173, Samara
  - saratov state medical /ID# 163130, Saratov
  - Yaroslavl Regional Clinic Hosp /ID# 162172, Yaroslavl
- South Africa (2):
  - Netcare Pretoria East Hospital /ID# 157373, Pretoria, Gauteng
  - Tshwane District Hospital /ID# 157361, Pretoria, Gauteng
- South Korea (4):
  - Pusan National University Hosp /ID# 158725, Busan, Busan Gwang Yeogsi
  - Chungnam National University Hospital /ID# 158726, Junggu, Daejeon Gwang Yeogsi
  - Cath Univ Seoul St Mary's Hosp /ID# 158724, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 162253, Seoul
- Spain (2):
  - Hospital Universitario y Politecnico La Fe /ID# 161181, Valencia, Valenciana
  - Hospital Infanta Leonor /ID# 161180, Madrid
- Taiwan (3):
  - National Taiwan Univ Hosp /ID# 162781, Taipei City, Taipei
  - Tri-Service General Hospital /ID# 161683, Taipei City, Taipei
  - Kaohsiung Medical University /ID# 161693, Kaohsiung City
- United Kingdom (3):
  - Heartlands Hospital /ID# 163534, Birmingham
  - University Hospital of Wales /ID# 162726, Cardiff
  - Northwick Park Hospital /ID# 162727, Harrow

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Wei AH, Montesinos P, Ivanov V, DiNardo CD, Novak J, Laribi K, Kim I, Stevens DA, Fiedler W, Pagoni M, Samoilova O, Hu Y, Anagnostopoulos A, Bergeron J, Hou JZ, Murthy V, Yamauchi T, McDonald A, Chyla B, Gopalakrishnan S, Jiang Q, Mendes W, Hayslip J, Panayiotidis P. Venetoclax plus LDAC for newly diagnosed AML ineligible for intensive chemotherapy: a phase 3 randomized placebo-controlled trial. Blood. 2020 Jun 11;135(24):2137-2145. doi: 10.1182/blood.2020004856. PMID 32219442
- [Derived] Wei AH, Panayiotidis P, Montesinos P, Laribi K, Ivanov V, Kim I, Novak J, Champion R, Fiedler W, Pagoni M, Bergeron J, Ting SB, Hou JZ, Yamauchi T, Wang J, Strickland SA, Savona MR, Lin TL, Enjeti AK, Tiong IS, Lee S, Roboz GJ, Popovic R, Jiang Q, Liu Z, Sun Y, Mendes WL, Chyla B, DiNardo CD. Risk stratification of low-dose cytarabine and venetoclax in patients with AML ineligible for intensive chemotherapy. Blood Adv. 2025 Nov 21:bloodadvances.2025017083. doi: 10.1182/bloodadvances.2025017083. Online ahead of print. PMID 41269778
- [Derived] Badawi M, Chen X, Marroum P, Suleiman AA, Mensing S, Koenigsdorfer A, Schiele JT, Palenski T, Samineni D, Hoffman D, Menon R, Salem AH. Bioavailability Evaluation of Venetoclax Lower-Strength Tablets and Oral Powder Formulations to Establish Interchangeability with the 100 mg Tablet. Clin Drug Investig. 2022 Aug;42(8):657-668. doi: 10.1007/s40261-022-01172-4. Epub 2022 Jul 13. PMID 35829925
- [Derived] Wei AH, Panayiotidis P, Montesinos P, Laribi K, Ivanov V, Kim I, Novak J, Stevens DA, Fiedler W, Pagoni M, Bergeron J, Ting SB, Hou JZ, Anagnostopoulos A, McDonald A, Murthy V, Yamauchi T, Wang J, Chyla B, Sun Y, Jiang Q, Mendes W, Hayslip J, DiNardo CD. 6-month follow-up of VIALE-C demonstrates improved and durable efficacy in patients with untreated AML ineligible for intensive chemotherapy (141/150). Blood Cancer J. 2021 Oct 1;11(10):163. doi: 10.1038/s41408-021-00555-8. PMID 34599139
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 76 sites globally. The study is currently ongoing; the results reported below include the primary analysis for efficacy which was conducted after 133 deaths occurred (data cut-off date of 15 February 2019), and an unplanned 6-month follow-up update for overall survival and safety (15 August 2019 cut-off date).
Pre-assignment Details: Participants with acute myeloid leukemia (AML) were randomized to one of two treatment arms in a 1:2 ratio (placebo + low-dose cytarabine [LDAC] or venetoclax + LDAC). Randomization was stratified by AML status (secondary, de novo), age (18 - < 75, ≥ 75) and region (United States [US], European Union [EU], China, Japan, rest of world).
Groups:
- Placebo + Low Dose Cytarabine (LDAC): Participants received matching placebo to venetoclax orally once a day (QD) plus cytarabine 20 mg/m² subcutaneously on Days 1 to 10 of each 28-day cycle.
  Participants continued treatment until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation were met.
- Venetoclax + Low Dose Cytarabine (LDAC): Participants received venetoclax 600 mg orally once a day plus cytarabine 20 mg/m² subcutaneously on Days 1 to 10 of each 28-day cycle.
  Participants continued treatment until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation were met.
Period: Overall Study
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Started | 68 | 143
Received Treatment | 68 | 142
Completed (As of 15 August 2019) | 56 | 103
Not Completed | 12 | 40
Not completed — Ongoing | 12 | 40

BASELINE CHARACTERISTICS:
Groups:
- Placebo + Low Dose Cytarabine (LDAC): Participants received matching placebo to venetoclax orally once a day (QD) plus cytarabine 20 mg/m² subcutaneously on Days 1 to 10 of each 28-day cycle.
- Venetoclax + Low Dose Cytarabine (LDAC): Participants received venetoclax 600 mg orally once a day plus cytarabine 20 mg/m² subcutaneously on Days 1 to 10 of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC) | Total
Number analyzed (Participants) | 68 | 143 | 211
Age, Continuous [Median (Full Range); unit: years] | 76.0 [41.0 to 88.0] | 76.0 [36.0 to 93.0] | 76.0 [36.0 to 93.0]
Age, Customized [Count of Participants; unit: Participants]
  18 to < 65 years | 9 | 11 | 20
  65 to < 75 years | 19 | 50 | 69
  ≥ 75 years | 40 | 82 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 65 | 94
  Male | 39 | 78 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 102 | 149
  Black or African American | 1 | 2 | 3
  Asian | 20 | 39 | 59
Region [Count of Participants; unit: Participants] — Rest of World includes Australia, Brazil, Canada, New Zealand, Puerto Rico, Russia, South Africa, South Korea, and Taiwan.
  Participants
    United States | 6 | 13 | 19
    European Union | 26 | 56 | 82
    China | 6 | 9 | 15
    Japan | 9 | 18 | 27
    Rest of World | 21 | 47 | 68
AML Status [Count of Participants; unit: Participants]
  De novo | 45 | 85 | 130
  Secondary | 23 | 58 | 81

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death. Participants who had not died were censored at the date they were last known to be alive on or before the cutoff date. Overall survival was analyzed using Kaplan-Meier methodology.
Time Frame: From randomization until the primary analysis cut-off date of February 15 2019; the median follow-up time was 12.0 months (range: 0.2-17.0) in the placebo arm and 12.0 months (range: 0.1-17.6) in the venetoclax arm.
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
months | 4.1 [3.1 to 8.8] | 7.2 [5.6 to 10.1]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.114, Log Rank; Log-rank test stratified by AML status (de novo, secondary) and age (18 - < 75, ≥ 75); Hazard Ratio (HR) = 0.749, 95% CI 2-sided [0.524 to 1.071] — The hazard ratio was estimated using the Cox proportional hazards model, stratified by AML status (de novo, secondary) and age (18 - < 75, ≥ 75)
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.103, Log Rank; Unstratified analysis; Hazard Ratio (HR) = 0.743, 95% CI 2-sided [0.521 to 1.061] — The hazard ratio was estimated using the Cox proportional hazards model

2. Secondary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Incomplete Blood Count Recovery (CR + CRi)
Description: The composite complete remission rate is defined as the percentage of participants with complete remission (CR) or complete remission with incomplete blood count recovery (CRi) at any time during the study as assessed by the investigator. Response was based on physical examination, bone marrow results and hematology values according to the revised guidelines by the International Working Group (IWG) for AML:
  CR: No morphologic evidence of AML and absolute neutrophil count (ANC) ≥ 10³/μL (1,000/μL), platelets ≥ 10⁵/μL (100,000/μL), red blood cell (RBC) transfusion independence, and bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  CRi: All criteria as CR except for residual neutropenia < 10³/μL or thrombocytopenia < 10⁵/μL. If all criteria for CR are met except RBC transfusion independence, the CRi criteria are met.
  Participants who had no IWG disease assessments were considered to be non-responders.
Time Frame: Response was assessed at the end of Cycle 1 and every 3 cycles thereafter to the end of treatment. Median treatment duration at the 15 February 2019 cut-off date was 1.7 months (range: 0.1-14.2) and 3.9 months (range: 0.0-17.1) in each group respectively.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 13.2 [6.2 to 23.6] | 47.6 [39.1 to 56.1]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary)
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Fisher Exact

3. Secondary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Partial Hematologic Recovery (CR + CRh)
Description: The percentage of participants who achieved a complete remission (CR) or complete remission with partial hematologic recovery (CRh) at any time point during the study assessed by the investigator.
  CR is defined according to the revised guidelines by the IWG for AML as no morphologic evidence of AML, ANC count ≥ 10³/μL, platelets ≥ 10⁵/μL, RBC transfusion independence, and bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  CRh is a derived response based on bone marrow blast and hematology lab values, achieved when the following criteria are met:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count of > 0.5 × 10³/μL and
  * Peripheral blood platelet count of > 0.5 × 10⁵/μL and
  * A 1 week platelet transfusion-free period prior to the hematology lab collection.
  Participants with no disease assessments were considered to be non-responders.
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 14.7 [7.3 to 25.4] | 46.9 [38.5 to 55.4]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary)
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Fisher Exact

4. Secondary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Incomplete Blood Count Recovery (CR + CRi) by Initiation of Cycle 2
Description: The composite complete remission rate is defined as the percentage of participants with complete remission (CR) or complete remission with incomplete blood count recovery (CRi) before initiation of Cycle 2, assessed by the investigator. Response was based on physical examination, bone marrow results and hematology values according to the revised guidelines by the IWG for AML:
  CR: No morphologic evidence of AML and absolute neutrophil count ≥ 10³/μL, platelets ≥ 10⁵/μL, red cell transfusion independence, and bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  CRi: All criteria as CR except for residual neutropenia < 10³/μL or thrombocytopenia < 10⁵/μL. If all criteria for CR are met except for RBC transfusion independence, CRi criteria are met.
  Participants who had no IWG disease assessments were considered to be non-responders.
Time Frame: Cycle 1, 28 days
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 2.9 [0.4 to 10.2] | 34.3 [26.5 to 42.7]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary)
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Fisher Exact

5. Secondary Outcome: Percentage of Participants With Complete Remission and Complete Remission With Partial Hematologic Recovery (CR + CRh) by Initiation of Cycle 2
Description: The percentage of participants who achieved a complete remission (CR) or complete remission with partial hematologic recovery (CRh) before initiation of Cycle 2 assessed by the investigator.
  CR is defined according to the revised guidelines by the IWG for AML as no morphologic evidence of AML, ANC count ≥ 10³/μL, platelets ≥ 10⁵/μL, RBC transfusion independence, and bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  CRh is a derived response based on bone marrow blast and hematology lab values, achieved when when the following criteria are met:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count of > 0.5 × 10³/μL and
  * Peripheral blood platelet count of > 0.5 × 10⁵/μL and
  * A 1-week platelet transfusion-free period prior to the hematology lab collection.
  Participants with no disease assessments were considered to be non-responders.
Time Frame: Cycle 1, 28 days
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 4.4 [0.9 to 12.4] | 30.8 [23.3 to 39.0]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary)
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Fisher Exact

6. Secondary Outcome: Percentage of Participants With Complete Remission
Description: The complete remission rate is defined as the percentage of participants with complete remission (CR) at any time during the study as assessed by the investigator. Response was based on physical examination, bone marrow results and hematology values according to the revised guidelines by the International Working Group (IWG) for AML. CR is defined as no morphologic evidence of AML and absolute neutrophil count ≥ 10³/μL, platelets ≥ 10⁵/μL, red blood cell transfusion independence, and bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  Participants who had no IWG disease assessments were considered to be non-responders.
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 7.4 [2.4 to 16.3] | 27.3 [20.2 to 35.3]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary)
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Fisher Exact

7. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form (SF) 7a
Description: PROMIS Fatigue SF 7a is a seven-item questionnaire that assesses the impact and experience of fatigue over the past 7 days. All questions employ the following five response options: 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, and 5 = Always. The PROMIS Fatigue 7a score is calculated as a T-score, which is a standardized score with a mean of 50 (based on the average for the United States general population) and a standard deviation (SD) of 10. Higher scores indicate higher levels of fatigue. A decrease in score (negative change from Baseline) indicates improvement in fatigue; the minimum important difference used in this study was 3 points.
Time Frame: Baseline and Day 1 of Cycles 3, 5, 7, and 9
Population: Full analysis set with available data at baseline and each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 60 | 127
score on a scale
  Cycle 3 Day 1: number analyzed (Participants) | 22 | 69
  Cycle 3 Day 1 | 1.567 (1.855) | -2.940 (1.093)
  Cycle 5 Day 1: number analyzed (Participants) | 12 | 40
  Cycle 5 Day 1 | -0.336 (2.307) | -5.259 (1.308)
  Cycle 7 Day 1: number analyzed (Participants) | 12 | 36
  Cycle 7 Day 1 | -3.818 (2.314) | -4.625 (1.354)
  Cycle 9 day 1: number analyzed (Participants) | 7 | 22
  Cycle 9 day 1 | -3.453 (2.811) | -5.101 (1.606)
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Cycle 3, Day 1; Test type: Other; LS Mean Difference = -4.507, 95% CI 2-sided [-8.60 to -0.41], Standard Error of Mean 2.068 — A linear mixed-effects regression model with a covariance structure including baseline score, stratification factors (age and AML status) treatment arm, visit, and treatment arm by visit interaction
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Cycle 5 Day 1; Test type: Other; LS Mean Difference = -4.923, 95% CI 2-sided [-10.03 to 0.19], Standard Error of Mean 2.580 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Cycle 7 Day 1; Test type: Other; LS Mean Difference = -0.807, 95% CI 2-sided [-5.98 to 4.36], Standard Error of Mean 2.609 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Cycle 9 day 1; Test type: Other; LS Mean Difference = -1.648, 95% CI 2-sided [-7.94 to 4.64], Standard Error of Mean 3.176 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); A linear mixed effects regression model with a variable covariance structure was fitted to the longitudinal data (considering all time points) to test for differences between treatment arms; Test type: Superiority; p = 0.126, Linear Mixed Effects Regression Model; Model included AML status (de novo vs. secondary), age (18-< 75 vs. ≥ 75), treatment arm, time, and treatment arm by time interaction as fixed factors

8. Secondary Outcome: Change From Baseline in Global Health Status / Quality of Life
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core (EORTC QLQ-C30) consists of a Global Health Status/Quality of Life (GHS/QoL) scale, a Financial Difficulties scale, 5 functional scales (Cognitive, Social, Physical, Emotional, and Role Functioning), and 8 symptom scales/items (Fatigue, Insomnia, Appetite Loss, Pain, Constipation, Diarrhea, Dyspnea, and Nausea and Vomiting).
  The GHS/QoL scale includes 2 questions in which participants were asked to rate their overall health and overall quality of life during the past week on a scale from 1 (very poor) to 7 (excellent). The 2 scores were averaged and transformed to a scale from 0 to 100, where a high score represents a high QoL. A positive change from baseline indicates better quality of life.
Time Frame: Baseline and Day 1 of Cycles 3, 5, 7, and 9
Population: Full analysis set with available data at Baseline and each time point
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 59 | 127
scores on a scale
  Cycle 3 Day 1: number analyzed (Participants) | 22 | 69
  Cycle 3 Day 1 | 1.941 (4.126) | 4.857 (2.413)
  Cycle 5 Day 1: number analyzed (Participants) | 12 | 40
  Cycle 5 Day 1 | 2.627 (5.047) | 16.015 (2.853)
  Cycle 7 Day 1: number analyzed (Participants) | 12 | 36
  Cycle 7 Day 1 | 3.481 (5.337) | 10.599 (3.092)
  Cycle 9 day 1: number analyzed (Participants) | 7 | 22
  Cycle 9 day 1 | 6.918 (6.642) | 13.299 (3.772)
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Cycle 3 Day 1; Test type: Other; LS Mean Difference = 2.917, 95% CI 2-sided [-6.23 to 12.06], Standard Error of Mean 4.617 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Cycle 5 Day 1; Test type: Other; LS Mean Difference = 13.388, 95% CI 2-sided [2.18 to 24.59], Standard Error of Mean 5.659 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Cycle 7 Day 1; Test type: Other; LS Mean Difference = 7.119, 95% CI 2-sided [-4.83 to 19.06], Standard Error of Mean 6.031 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Cycle 9 Day 1; Test type: Other; LS Mean Difference = 6.381, 95% CI 2-sided [-8.49 to 21.26], Standard Error of Mean 7.511 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); [analysis description as in outcome 7, analysis 5]; Test type: Superiority; p = 0.085, Linear Mixed Effects Regression Model; [statistical method as in outcome 7, analysis 5]

9. Secondary Outcome: Event-free Survival (EFS)
Description: Event-free survival is defined as the time from randomization to the date of progressive disease (PD), confirmed morphologic relapse from CR or CRi, treatment failure (failure to achieve CR, CRi or morphologic leukemia free state (MLFS) after at least 6 cycles of study treatment), or death from any cause, assessed by the investigator according to the modified IWG criteria.
  PD:
  * > 50% increase in marrow blasts (minimum 15% increase required if blasts < 30% at baseline); or persistent marrow blast > 70% for ≥ 3 months; without at least a 100% improvement in ANC to an absolute level > 0.5 × 10⁹/L, and/or platelets to > 50 × 10⁹/L non-transfused; or
  * 50% increase in peripheral blasts to > 25 × 10⁹/L; or
  * New extramedullary disease
  Participants with no events prior to the cut-off date were censored at their last assessment date; participants with no events prior to post-treatment therapy initiated before the cut-off date were censored on the start date of post-treatment therapy.
Time Frame: From randomization until the primary analysis cut-off date of February 15, 2019; the median follow-up time was 12.0 months (range: 0.2-17.0) in the placebo arm and 12.0 months (range: 0.1-17.6) in the venetoclax arm.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
months | 2.0 [1.6 to 3.1] | 4.7 [3.7 to 6.4]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.002, Log Rank; Log-rank test stratified by AML status (de novo, secondary) and age (18 - < 75, ≥ 75); Hazard Ratio (HR) = 0.583, 95% CI 2-sided [0.416 to 0.817] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.003, Log Rank; Unstratified analysis; Hazard Ratio (HR) = 0.601, 95% CI 2-sided [0.430 to 0.839] — The hazard ratio was estimated using the Cox proportional hazards model

10. Secondary Outcome: Percentage of Participants With Post Baseline Red Blood Cell (RBC) Transfusion Independence
Description: The post baseline red blood cell (RBC) transfusion independence rate was calculated as the percentage of participants who achieved RBC transfusion independence post baseline. RBC transfusion independence is defined as a period of at least 56 consecutive days with no RBC transfusion after the first dose of study drug and on or before the last dose of study drug plus 30 days, or disease progression, or confirmed morphological relapse, or death, or the data cut-off date, whichever occurred earlier.
Time Frame: From first dose of study drug until 30 days after last dose up to the data cut-off date of 15 February 2019; Median time on treatment was 1.7 months (range: 0.1-14.2) in the placebo arm and 3.9 months (range: 0.0-17.1) in the venetoclax arm.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 17.6 [9.5 to 28.8] | 40.6 [32.4 to 49.1]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary); Treatment Difference = 22.9, 95% CI 2-sided [10.8 to 35.0] — Treatment difference = Venetoclax - Placebo
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p < 0.001, Fisher Exact

11. Secondary Outcome: Percentage of Participants With Post Baseline Platelet Transfusion Independence
Description: The post baseline platelet transfusion independence rate was calculated as the percentage of participants who achieved platelet transfusion independence post Baseline. Platelet transfusion independence is defined as a period of at least 56 consecutive days with no platelet transfusion after the first dose of study drug and on or before the last dose of study drug plus 30 days, or disease progression, or confirmed morphological relapse, or death, or the data cut--off date, whichever occurred earlier.
Time Frame: as for outcome 10
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 32.4 [21.5 to 44.8] | 47.6 [39.1 to 56.1]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.040, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary); Treatment Difference = 15.2, 95% CI 2-sided [1.4 to 29.0] — Treatment difference = Venetoclax - Placebo
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.039, Fisher Exact

12. Secondary Outcome: Percentage of Participants With RBC Transfusion Independence Among Those Who Were Transfusion Dependent at Baseline
Description: The rate of conversion was calculated as the percentage of participants who were post-baseline RBC transfusion independent among participants who had an RBC transfusion within 8 weeks prior to the first dose of study drug (i.e. were transfusion dependent at Baseline). RBC transfusion independence is defined as a period of at least 56 days with no RBC transfusion after the first dose of study drug and on or before the last dose of study drug plus 30 days, or disease progression, or confirmed morphological relapse, or death, or the data cut-off date, whichever occurred earlier.
Time Frame: as for outcome 10
Population: Full analysis set participants who were RBC transfusion-dependent at Baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 53 | 104
percentage of participants | 15.1 [6.7 to 27.6] | 37.5 [28.2 to 47.5]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; Treatment Difference = 22.4, 95% CI 2-sided [9.0 to 35.8]

13. Secondary Outcome: Percentage of Participants With Platelet Transfusion Independence Among Those Who Were Transfusion Dependent at Baseline
Description: The rate of conversion was calculated as the percentage of participants who were post-baseline platelet transfusion independent among participants who had a platelet transfusion within 8 weeks prior to the first dose of study drug (i.e. were transfusion dependent at Baseline). Platelet transfusion independence is defined as a period of at least 56 days with no platelet transfusion after the first dose of study drug and on or before the last dose of study drug plus 30 days, or disease progression, or confirmed morphological relapse, or death, or the data cut-off date, whichever occurred earlier.
Time Frame: as for outcome 10
Population: Full analysis participants who were platelet transfusion dependent at Baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 24 | 53
percentage of participants | 12.5 [2.7 to 32.4] | 30.2 [18.3 to 44.3]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; Slope = 17.7, 95% CI 2-sided [-0.4 to 35.8]

14. Secondary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Incomplete Blood Count Recovery (CR + CRi) and Minimal Residual Disease (MRD) Response
Description: The percentage of participants with complete remission or complete remission with incomplete blood count recovery AND minimal residual disease (MRD) as assessed by the investigator. Response was based on the modified IWG response criteria for AML:
  CR: No morphologic evidence of AML and ANC ≥ 10³/μL, platelets ≥ 10⁵/μL, red blood cell (RBC) transfusion independence, and bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  CRi: All criteria as CR except for residual neutropenia < 10³/μL or thrombocytopenia < 10⁵/μL. If all criteria for CR are met except RBC transfusion independence, CRi criteria are met.
  MRD response (at lowest-point MRD value) was defined as having less than 10-³ residual blasts per leukocyte measured in the bone marrow, per European LeukemiaNet (ELN) recommendations.
  Participants who had no disease or MRD assessments were considered to be non-responders.
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 1.5 [0.0 to 7.9] | 5.6 [2.4 to 10.7]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.162, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary)
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.277, Fisher Exact

15. Secondary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Partial Hematologic Recovery (CR + CRh) and Minimal Residual Disease (MRD) Response
Description: The percentage of participants with complete remission or complete remission with partial hematologic recovery (CRh) AND MRD response as assessed by the investigator.
  CR is defined according to the modified IWG response criteria for AML as no morphologic evidence of AML, ANC ≥ 10³/μL, platelets ≥ 10⁵/μL, RBC transfusion independence, and bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  CRh is achieved when the following criteria are met:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count of > 0.5 × 10³/μL and
  * Peripheral blood platelet count of > 0.5 × 10⁵/μL and
  * A 1 week platelet transfusion-free period prior to the hematology lab collection.
  MRD response (at lowest-point MRD value) was defined as less than 10-³ residual blasts per leukocyte measured in the bone marrow, per ELN recommendations.
  Participants who had no disease or MRD assessments were considered to be non-responders.
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants | 1.5 [0.0 to 7.9] | 5.6 [2.4 to 10.7]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.162, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (18 - < 75, ≥ 75) and AML status (de novo, secondary)
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Superiority; p = 0.277, Fisher Exact

16. Secondary Outcome: Overall Survival (OS) by Mutation Subgroups
Description: Overall survival is defined as the time from the date of randomization to the date of death. Participants who had not died were censored at the date they were last known to be alive on or before the cutoff date. Overall survival was analyzed using Kaplan-Meier methodology.
  Overall survival was analyzed in participants with the following molecular markers:
  * Isocitrate dehydrogenase 1 and 2 (IDH1/2) mutation
  * FMS (Feline McDonough Sarcoma)-like tyrosine kinase 3 (FLT3) mutation
Time Frame: as for outcome 9
Population: The full analysis set; participants in each mutation subgroup
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
months
  IDH1/2 mutation: number analyzed (Participants) | 12 | 21
  IDH1/2 mutation | 9.0 [2.2 to NA] — Could not be calculated due to the low number of events | 10.8 [4.2 to NA] — Could not be calculated due to the low number of events
  FLT3 mutation: number analyzed (Participants) | 9 | 20
  FLT3 mutation | 9.8 [0.9 to NA] — Could not be calculated due to the low number of events | 5.9 [1.6 to 10.9]

17. Secondary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Incomplete Blood Count Recovery (CR + CRi) by Mutation Subgroup
Description: Response was based on physical examination, bone marrow results and hematology values according to the revised guidelines by the IWG for AML:
  CR: No morphologic evidence of AML and ANC ≥ 10³/μL, platelets ≥ 10⁵/μL, RBC transfusion independence, and bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  CRi: All criteria as CR except for residual neutropenia < 10³/μL or thrombocytopenia < 10⁵/μL. If all criteria for CR are met except RBC transfusion independence, CRi criteria is met.
  Participants who had no IWG disease assessments were considered to be non-responders.
  Response was analyzed in participants with the following mutations:
  * Isocitrate dehydrogenase 1 and 2 (IDH1/2) mutation
  * FMS-like tyrosine kinase 3 (FLT3) mutation
Time Frame: as for outcome 2
Population: Full analysis set participants in each mutation subgroup
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants
  IDH1/2 mutation: number analyzed (Participants) | 12 | 21
  IDH1/2 mutation | 33.3 | 57.1
  FLT3 mutation: number analyzed (Participants) | 9 | 20
  FLT3 mutation | 44.4 | 45.0

18. Secondary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Partial Hematologic Recovery (CR + CRh) by Mutation Subgroup
Description: The percentage of participants who achieved a complete remission or complete remission with partial hematologic recovery assessed by the investigator for participants with the following mutations:
  * Isocitrate dehydrogenase 1 and 2 (IDH1/2) mutation
  * FMS-like tyrosine kinase 3 (FLT3) mutation
  CR is defined according to the modified IWG criteria for AML as no morphologic evidence of AML, ANC ≥ 10³/μL, platelets ≥ 10⁵/μL, RBC transfusion independence, bone marrow with < 5% blasts, absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
  CRh is achieved when the following criteria are met:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count > 0.5 × 10³/μL and
  * Peripheral blood platelet count > 0.5 × 10⁵/μL and
  * A 1 week platelet transfusion-free period prior to hematology lab collection. Participants with no disease assessments were considered non-responders
Time Frame: as for outcome 2
Population: Full analysis set participants in each mutation subgroup
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
percentage of participants
  IDH1/2 mutation: number analyzed (Participants) | 12 | 21
  IDH1/2 mutation | 33.3 | 57.1
  FLT3 mutation: number analyzed (Participants) | 9 | 20
  FLT3 mutation | 44.4 | 45.0

19. Post Hoc Outcome: Overall Survival After an Additional 6-Months Follow-up
Description: as for outcome 1
Time Frame: From randomization until the 6-month follow-up analysis cut-off date of August 15, 2019; the median follow-up time was 17.7 months (range: 0.2-20.8) in the placebo arm and 17.5 months (range: 0.1-23.5) in the venetoclax arm.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
Number analyzed (Participants) | 68 | 143
months | 4.1 [3.1 to 8.1] | 8.4 [5.9 to 10.1]
Statistical Analysis 1: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Other; p = 0.040, Log Rank; Log-rank test stratified by AML status (de novo, secondary) and age (18 - < 75, ≥ 75); Hazard Ratio (HR) = 0.704, 95% CI 2-sided [0.503 to 0.985] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo + Low Dose Cytarabine (LDAC) vs Venetoclax + Low Dose Cytarabine (LDAC); Test type: Other; p = 0.049, Log Rank; Unstratified analysis; Hazard Ratio (HR) = 0.717, 95% CI 2-sided [0.514 to 1.000] — The hazard ratio was estimated using the Cox proportional hazards model

ADVERSE EVENTS:
Time Frame: All-cause mortality includes all deaths up to the data cut-off date of 15 August 2019; median time on study was 17.7 months (range: 0.2-20.8) in the placebo arm and 17.5 months (range: 0.1-23.5) in the venetoclax arm. Adverse events are reported from the first dose of study drug up to 30 days after the last dose, to the data cut-off date of 15 August 2019; median duration of treatment was 1.7 months (range: 0.1-20.2) in the placebo arm and 4.1 months (range: 0.0-23.5) in the venetoclax arm.
Arm/Group | Placebo + Low Dose Cytarabine (LDAC) | Venetoclax + Low Dose Cytarabine (LDAC)
All-Cause Mortality (participants affected / at risk) | 54/68 | 99/142
Serious Adverse Events (participants affected / at risk) | 42/68 | 95/142
Other Adverse Events (participants affected / at risk) | 65/68 | 135/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Low Dose Cytarabine (LDAC) (N=68) | Venetoclax + Low Dose Cytarabine (LDAC) (N=142)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 12 (14) | 24 (32)
HYPERLEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 7 (8)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 3 (3) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 4 (5)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1)
EYELID HAEMATOMA (Eye disorders) | 0 (0) | 1 (1)
EYELID OEDEMA (Eye disorders) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (2) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (2)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (4)
DEATH (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 5 (7) | 3 (3)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 2 (2)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
ABSCESS NECK (Infections and infestations) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
ASPERGILLUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 (1) | 1 (1)
CANDIDA SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 4 (4)
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 2 (2)
ENTEROCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
EXTERNAL EAR CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
KLEBSIELLA INFECTION (Infections and infestations) | 1 (1) | 1 (1)
KLEBSIELLA SEPSIS (Infections and infestations) | 2 (2) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 1 (2) | 0 (0)
LUNG INFECTION (Infections and infestations) | 2 (2) | 4 (4)
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 1 (1) | 0 (0)
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
MUCORMYCOSIS (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 3 (3)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
PAROTITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 7 (7) | 20 (24)
PNEUMONIA FUNGAL (Infections and infestations) | 0 (0) | 2 (2)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
PSOAS ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY MYCOSIS (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 4 (4) | 8 (8)
SEPTIC SHOCK (Infections and infestations) | 4 (4) | 5 (5)
SERRATIA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2 (2) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (4)
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRAUMATIC HAEMOTHORAX (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (4)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (4)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TUMOUR ASSOCIATED FEVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 1 (1)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
ORTHOSTATIC INTOLERANCE (Nervous system disorders) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 2 (2)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Low Dose Cytarabine (LDAC) (N=68) | Venetoclax + Low Dose Cytarabine (LDAC) (N=142)
ANAEMIA (Blood and lymphatic system disorders) | 15 (17) | 37 (60)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 8 (11) | 22 (24)
LEUKOPENIA (Blood and lymphatic system disorders) | 5 (6) | 13 (17)
NEUTROPENIA (Blood and lymphatic system disorders) | 12 (14) | 65 (130)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 25 (37) | 58 (117)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 17 (17)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 9 (11)
CONSTIPATION (Gastrointestinal disorders) | 22 (25) | 29 (38)
DIARRHOEA (Gastrointestinal disorders) | 12 (15) | 46 (70)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 9 (11)
NAUSEA (Gastrointestinal disorders) | 21 (27) | 61 (95)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 14 (15)
VOMITING (Gastrointestinal disorders) | 10 (10) | 41 (59)
ASTHENIA (General disorders) | 8 (10) | 17 (20)
FATIGUE (General disorders) | 10 (10) | 22 (27)
MALAISE (General disorders) | 4 (4) | 4 (8)
OEDEMA PERIPHERAL (General disorders) | 14 (15) | 20 (27)
PYREXIA (General disorders) | 8 (10) | 22 (26)
ORAL HERPES (Infections and infestations) | 1 (1) | 9 (9)
PNEUMONIA (Infections and infestations) | 4 (6) | 11 (12)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 13 (15)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5) | 9 (14)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 12 (15)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 16 (17)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (5) | 9 (13)
PLATELET COUNT DECREASED (Investigations) | 3 (7) | 8 (18)
WEIGHT DECREASED (Investigations) | 2 (3) | 14 (18)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 4 (8) | 9 (22)
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 (14) | 30 (35)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 5 (5) | 6 (9)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 (3) | 11 (12)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 9 (11) | 9 (11)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 8 (10) | 13 (14)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 17 (24) | 44 (63)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 6 (6) | 13 (14)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 7 (7) | 8 (8)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 4 (4) | 5 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 12 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (6) | 9 (9)
DIZZINESS (Nervous system disorders) | 1 (1) | 12 (14)
HEADACHE (Nervous system disorders) | 3 (3) | 20 (28)
CONFUSIONAL STATE (Psychiatric disorders) | 5 (5) | 3 (3)
INSOMNIA (Psychiatric disorders) | 9 (9) | 20 (20)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 5 (6) | 6 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 14 (17)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 11 (14)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 15 (20)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (8)
RASH (Skin and subcutaneous tissue disorders) | 5 (7) | 10 (13)
HYPERTENSION (Vascular disorders) | 7 (8) | 14 (14)
HYPOTENSION (Vascular disorders) | 2 (3) | 13 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT03069352/Prot_001.pdf
  • Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT03069352/SAP_000.pdf